CLINICAL TRIAL: NCT03843411
Title: Mini-fluid Challenge as a Predictor of Fluid Response for Pneumoperitoneum Patient
Status: Withdrawn | Type: Observational
Why Stopped: no funding
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 181239
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Anesthesia
Keywords: mini-fluid challenge

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate whether the change of stroke volume index(△SVI) induced by the rapid mini-fluid administration can predict fluid responsiveness in patients with pneumoperitoneum

DETAILED DESCRIPTION:
Perioperative fluid management is significant important during surgery. The current trend tends to use goal-directed fluid therapy in surgery. Goal-directed fluid therapy refers to continuous monitoring of hemodynamic parameters during surgery and managing more accurate fluid administration based on the data obtained while promoting optimal tissue perfusion. Define fluid responsiveness with the hemodynamic parameters as to whether the cardiac output can be significantly increased after administration of fluid. Therefore, the advantage of predicting fluid responsiveness is that it can optimize the cardiac output and tissue perfusion while avoiding administering unnecessary fluid to patients.

The purpose of this study is to evaluate whether the change of stroke volume index(△SVI) induced by the rapid mini-fluid administration can predict fluid responsiveness in patients with pneumoperitoneum.

ELIGIBILITY:
Inclusion Criteria:

* receive operation that required pneumoperitoneum and FloTrac monitoring
* ASA 1~3
* age between 20 to 70 year old

Exclusion Criteria:

* patient who cannot understand the process and aim of the study
* patient with arrhythmia
* poor heart function(LVEF<50%, severe valvular disease, CAD)
* CKD
* pregnant patient
* patients allergic to voluven

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: receive operation that required pneumoperitoneum and FloTrac monitoring
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
change of stroke volume index | 1 hours
  record stroke volume index before and after mini-fluid challenge